CLINICAL TRIAL: NCT00303810
Title: Multicenter Therapy Optimizing Study for Treatment of Children and Adolescents With Intracranial Medulloblastoma / PNET and Ependymoma
Brief Title: Radiation Therapy and Combination Chemotherapy in Treating Young Patients With Medulloblastoma, Supratentorial Primitive Neuroectodermal Tumor, or Ependymoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000455572; GPOH-HIT-2000; EU-205105
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2009-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood infratentorial ependymoma; childhood supratentorial ependymoma; untreated childhood medulloblastoma; newly diagnosed childhood ependymoma; untreated childhood supratentorial primitive neuroectodermal tumor
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Carboplatin; Cisplatin; Cyclophosphamide; etoposide phosphate; Drug Therapy; Lomustine; Methotrexate; Thiotepa; Vincristine; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: cyclophosphamide
Drug: etoposide phosphate
Drug: high-dose chemotherapy
Drug: lomustine
Drug: methotrexate
Drug: thiotepa
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy in different ways and giving it together with more than one drug (combination chemotherapy) may kill more tumor cells. It is not yet known which radiation therapy and combination chemotherapy regimen is more effective in treating medulloblastoma, supratentorial primitive neuroectodermal tumor (PNET), or ependymoma.

PURPOSE: This clinical trial is studying six different radiation therapy and combination chemotherapy regimens to compare how well they work in treating young patients with medulloblastoma, PNET, or ependymoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare prognosis, using adapted risk stratification and quality control of diagnostic assessments and therapy, in pediatric patients with intracranial medulloblastoma, supratentorial primitive neuroectodermal tumor (PNET), or ependymoma treated with intensified chemotherapy and radiotherapy.
* Determine the effect of omission of radiotherapy, in terms of long-term sequelae, in young children with medulloblastoma and by hyperfractionation and reduction of radiotherapy in older children with medulloblastoma.
* Compare hyperfractionated radiotherapy with reduced-dose radiotherapy in older children with stage M0 medulloblastoma.

OUTLINE: This is a multi-protocol study. Patients are enrolled on 1 of 6 treatment protocols according to diagnosis and age at diagnosis.

* Protocol HIT-2000-AB4 (≥ 4 years old at diagnosis with nonmetastatic medulloblastoma)(phase III randomized controlled multicenter study): Patients are randomized to undergo hyperfractionated radiotherapy or conventional reduced-dose radiotherapy, followed by vincristine, lomustine, and cisplatin.
* Protocol HIT-2000-BIS4 (< 4 years old at diagnosis with nonmetastatic medulloblastoma): Patients receive 5 courses of cyclophosphamide, vincristine, methotrexate, carboplatin, etoposide phosphate, and intrathecal methotrexate. Patients with residual tumors after 3 courses undergo conventionally fractionated reduced-dose radiotherapy.
* Protocol MET-HIT-2000-AB4 (≥ 4 years old at diagnosis with metastatic medulloblastoma or supratentorial PNET): Patients receive combination chemotherapy as in HIT-2000-BIS4 for 2 courses. Patients then undergo hyperfractionated radiotherapy and receive combination chemotherapy as in HIT-2000-AB4. Patients with good response to combination chemotherapy (as in HIT-2000-BIS4) also receive high-dose chemotherapy.
* Protocol MET-HIT-2000-BIS4 (< 4 years old at diagnosis with metastatic medulloblastoma or supratentorial PNET): Patients receive 2-4 courses of carboplatin IV and etoposide phosphate IV continuously over 96 hours. Patients with partial or complete response also receive high-dose carboplatin, etoposide phosphate, cyclophosphamide, and thiotepa. Patients with residual tumor undergo conventional fractionated, reduced-dose radiotherapy.
* Protocol E-HIT-2000-AB4 (≥ 4 years old at diagnosis with intracranial ependymoma): Patients undergo local hyperfractionated radiotherapy. If histological grading shows WHO grade III tumor, patients also receive 5 courses of vincristine, cyclophosphamide, carboplatin, and etoposide phosphate.
* Protocol E-HIT-2000-BIS4 (< 4 years old at diagnosis with intracranial ependymoma): Patients receive 5 courses of cyclophosphamide, vincristine, methotrexate IV, carboplatin, and etoposide phosphate and then undergo conventional fractionated local radiotherapy.

PROJECTED ACCRUAL: A total of 567 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Medulloblastoma
  * Supratentorial primitive neuroectodermal tumor (PNET)
  * Ependymoma
* Intracranial tumor

  * No brain stem tumors
* No recurrent or relapsed tumors

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 567 (Actual)
Dates: Start 2001-01; Primary Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Rutkowski, MD, Study Chair — University Med. Center Hamburg, Dpt. of Pediatric Hematology and Oncology; Frank Deinlein, MD — Universitaets - Kinderklinik Wuerzburg
Locations (1):
- University Medical Center Hamburg - Eppendorf, Hamburg, Germany

REFERENCES:
- [Result] von Bueren AO, von Hoff K, Pietsch T, Gerber NU, Warmuth-Metz M, Deinlein F, Zwiener I, Faldum A, Fleischhack G, Benesch M, Krauss J, Kuehl J, Kortmann RD, Rutkowski S. Treatment of young children with localized medulloblastoma by chemotherapy alone: results of the prospective, multicenter trial HIT 2000 confirming the prognostic impact of histology. Neuro Oncol. 2011 Jun;13(6):669-79. doi: 10.1093/neuonc/nor025. PMID 21636711
- [Derived] Mynarek M, von Hoff K, Pietsch T, Ottensmeier H, Warmuth-Metz M, Bison B, Pfister S, Korshunov A, Sharma T, Jaeger N, Ryzhova M, Zheludkova O, Golanov A, Rushing EJ, Hasselblatt M, Koch A, Schuller U, von Deimling A, Sahm F, Sill M, Riemenschneider MJ, Dohmen H, Monoranu CM, Sommer C, Staszewski O, Mawrin C, Schittenhelm J, Bruck W, Filipski K, Hartmann C, Meinhardt M, Pietschmann K, Haberler C, Slavc I, Gerber NU, Grotzer M, Benesch M, Schlegel PG, Deinlein F, von Bueren AO, Friedrich C, Juhnke BO, Obrecht D, Fleischhack G, Kwiecien R, Faldum A, Kortmann RD, Kool M, Rutkowski S. Nonmetastatic Medulloblastoma of Early Childhood: Results From the Prospective Clinical Trial HIT-2000 and An Extended Validation Cohort. J Clin Oncol. 2020 Jun 20;38(18):2028-2040. doi: 10.1200/JCO.19.03057. Epub 2020 Apr 24. PMID 32330099
- [Derived] von Bueren AO, Kortmann RD, von Hoff K, Friedrich C, Mynarek M, Muller K, Goschzik T, Zur Muhlen A, Gerber N, Warmuth-Metz M, Soerensen N, Deinlein F, Benesch M, Zwiener I, Kwiecien R, Faldum A, Bode U, Fleischhack G, Hovestadt V, Kool M, Jones D, Northcott P, Kuehl J, Pfister S, Pietsch T, Rutkowski S. Treatment of Children and Adolescents With Metastatic Medulloblastoma and Prognostic Relevance of Clinical and Biologic Parameters. J Clin Oncol. 2016 Dec;34(34):4151-4160. doi: 10.1200/JCO.2016.67.2428. Epub 2016 Oct 31. PMID 27863192
- [Derived] Pompe RS, von Bueren AO, Mynarek M, von Hoff K, Friedrich C, Kwiecien R, Treulieb W, Lindow C, Deinlein F, Fleischhack G, Kuehl J, Rutkowski S. Intraventricular methotrexate as part of primary therapy for children with infant and/or metastatic medulloblastoma: Feasibility, acute toxicity and evidence for efficacy. Eur J Cancer. 2015 Nov;51(17):2634-42. doi: 10.1016/j.ejca.2015.08.009. Epub 2015 Sep 4. PMID 26346136
- [Derived] von Bueren AO, Friedrich C, von Hoff K, Kwiecien R, Muller K, Pietsch T, Warmuth-Metz M, Hau P, Benesch M, Kuehl J, Kortmann RD, Rutkowski S. Metastatic medulloblastoma in adults: outcome of patients treated according to the HIT2000 protocol. Eur J Cancer. 2015 Nov;51(16):2434-43. doi: 10.1016/j.ejca.2015.06.124. Epub 2015 Aug 5. PMID 26254812
- [Derived] Gerber NU, von Hoff K, Resch A, Ottensmeier H, Kwiecien R, Faldum A, Matuschek C, Hornung D, Bremer M, Benesch M, Pietsch T, Warmuth-Metz M, Kuehl J, Rutkowski S, Kortmann RD. Treatment of children with central nervous system primitive neuroectodermal tumors/pinealoblastomas in the prospective multicentric trial HIT 2000 using hyperfractionated radiation therapy followed by maintenance chemotherapy. Int J Radiat Oncol Biol Phys. 2014 Jul 15;89(4):863-71. doi: 10.1016/j.ijrobp.2014.04.017. PMID 24969797